CLINICAL TRIAL: NCT00391924
Title: Fatigue and General Well-Being in Patients With Systemic Lupus Erythematosus or Primary Sjögren's Syndrome: Effects of Dehydroepiandrosterone Administration
Brief Title: Dehydroepiandrosterone Administration in Women With Systemic Lupus Erythematosus or Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: University Medical Center Groningen (Other); Dutch Arthritis Association (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NR 98-2-301
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2006-10

CONDITIONS: Lupus Erythematosus, Systemic; Sjogren's Syndrome
Keywords: Dehydroepiandrosterone; Fatigue; Quality of life; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Bone mineral density
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Fatigue | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: Dehydroepiandrosterone

SUMMARY:
The purpose of the study is to examine whether dehydroepiandrosterone (DHEA) administration improves fatigue and general well-being in patients with systemic lupus erythematosus or primary Sjögren's syndrome

DETAILED DESCRIPTION:
Fatigue and reduced general well-being are frequent complaints in patients with the chronic autoimmune disorder systemic lupus erythematosus (SLE) or primary Sjögren's syndrome (pSS). Uncontrolled studies suggested that the administration of dehydroepiandrosterone (DHEA) may improve such complaints. The aim of our randomized double-blind placebo-controlled study is to examine the effect of daily oral 200 mg DHEA on fatigue, well-being, and functioning in women with SLE or pSS.

ELIGIBILITY:
Inclusion Criteria:

* pSS with a focus score >= 1 on minor salivary gland biopsy and fulfilling European classification criteria (Ann Rheum Dis 1996;55:116-21)
* SLE according to ACR classification criteria (Arthritis Rheum 1982;25:1271-7)
* Willingness to apply effective contraception (premenopausal women)
* Written informed consent.

Exclusion Criteria:

* Pregnancy
* Pregnancy wish
* Serum creatinine > 150 µmol/L
* Glucocorticoid use at a daily dose > 10 mg prednisone (or equivalent)
* Cyclophosphamide treatment in the preceding year
* Hyper- or hypothyroidism
* History of malignancy within the previous 5 years with exception of squamous or basal cell carcinoma of the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-05; Study Completion 2003-01

PRIMARY OUTCOMES:
General fatigue
Depressive mood
Mental well-being
Physical functioning
(all measures at baseline, after 3, 6, and 12 months of intake of study medication, and 6 months after cessation of medication intake)

SECONDARY OUTCOMES:
Self-reported pain,
Fibromyalgia tender points
Erythrocyte sedimentation rate
Hemoglobin
Serum Immunoglobulin-G
Self-reported ocular dryness (in pSS only)
Self-reported oral dryness (in pSS only)
Ocular tear production (in pSS only)
SLE disease activity index (in SLE only)
Bone mineral density (in SLE only)
Dose of glucocorticoids (in SLE only)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald HW Derksen, MD,PhD, Study Chair — UMC Utrecht
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Result] Hartkamp A, Geenen R, Godaert GL, Bijl M, Bijlsma JW, Derksen RH. The effect of dehydroepiandrosterone on lumbar spine bone mineral density in patients with quiescent systemic lupus erythematosus. Arthritis Rheum. 2004 Nov;50(11):3591-5. doi: 10.1002/art.20610. PMID 15529389
- [Result] Hartkamp A, Geenen R, Bijl M, Kruize AA, Godaert GL, Derksen RH. Serum cytokine levels related to multiple dimensions of fatigue in patients with primary Sjogren's syndrome. Ann Rheum Dis. 2004 Oct;63(10):1335-7. doi: 10.1136/ard.2003.011825. PMID 15361396
- [Derived] Hartkamp A, Geenen R, Godaert GL, Bijl M, Bijlsma JW, Derksen RH. Effects of dehydroepiandrosterone on fatigue and well-being in women with quiescent systemic lupus erythematosus: a randomised controlled trial. Ann Rheum Dis. 2010 Jun;69(6):1144-7. doi: 10.1136/ard.2009.117036. Epub 2009 Oct 22. PMID 19854713